CLINICAL TRIAL: NCT07050290
Title: Restoring Segmental Lordosis Via One Previous Posterior Approach After Failed Fusion at the Same Level for Degenerative Lumbar Disease
Brief Title: Restoring Segmental Lumbar Lordosis After Failed Previous Fusion at the Same Level
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: N.N. Priorov National Medical Research Center of Traumatology and Orthopedics (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NS12-04
Record Dates: First submitted 2025-06-25; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Failed Back Surgery Syndrome; Degeneration Lumbar Spine; Degenerative Spondylolisthesis; Sagittal Imbalance
Keywords: Lumbar fusion; segmental lordosis; revision spinal surgery; posterior approach
MeSH Terms: conditions — Failed Back Surgery Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cohort (Other): All patients will undergo restoring segmental lordosis via one previous posterior approach after failed fusion at the same level.
  Interventions: Procedure: Restoring segmental lordosis at the lumbar spine

INTERVENTIONS:
Procedure: Restoring segmental lordosis at the lumbar spine — All patients will undergo restoring segmental lordosis via one previous posterior approach after failed fusion at the same level.

SUMMARY:
The restoration of lumbar lordosis is mandatory during lumbar fusion surgery for degenerative disc disease, since not restoring lumbar lordosis adequately may adversely affect surgical outcomes and the patient's quality of life in the follow-up. Revision surgery to restore segmental lordosis at the level of previous spinal fusion is extremely difficult to do and its performance is usually inferior to that of primary surgery. Need to provide a surgical technique to restore segmental lordosis via a posterior approach, which is especially important after failed previous fusion at the same lumbar level.

ELIGIBILITY:
Inclusion Criteria:

* 1. Over 18 years' old;
* 2. Lumbar back pain with / without radicular leg pain (with / without neurological deficit) with / without neurogenic claudication, symptoms persisting for at least 3 months prior to surgery;
* 3. 1) Failed back lumbar fusion surgery at the same level or on an adjacent segment or 2) Symptomatic discopathy with loss of segmental lordosis at one of the levels L3-L4, L4-L5 or L5-S1, confirmed by MRI и Rg, with/without degenerative stenosis/spondylolisthesis
* 4. Need for a planned surgical procedure with a major extent of segmental lordosis restoration (more than 10°);
* 5. Given written informed consent;
* 6. Able and agree to fully comply with the clinical protocol and willing to adhere to follow-up schedule and requirements

Exclusion Criteria:

* 1. Interbody implants previously placed via non-posterior approach at the level of surgery (which cannot be removed through the posterior approach);
* 2. Complete interbody fusion after previous surgery at the level of surgery;
* 3. HU values of lumbar body vertebrae less than 120 HU;
* 4. Any contraindication or inability to undergo baseline and/or follow up MRI, CT or X-ray as required per protocol;
* 5. Back or non-radicular pain of unknown etiology;
* 6. History or presence of any other major neurological disease or condition that may interfere with the study assessments;
* 7. Previous enrollment in this study, current enrollment or plans to be enrolled in another study (in parallel to this study).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-06-25 (Actual); Primary Completion 2026-07-25 (Estimated); Study Completion 2027-07-25 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in lumbar balance parameters | 2 weeks postoperatively (or at day of hospital discharge)
  To observe the change from baseline in segmental lordosis at operated level by CT, in degrees

SECONDARY OUTCOMES:
Change from baseline in Numeric Pain Rating Scale | 2 weeks (or at day of hospital discharge), 3 months, 12 months postoperatively
  To observe the change of Numeric Pain Rating Scale as compared to baseline through follow-up terms (0 - no pain, 10 - unbearable pain)
Change from baseline in Oswestry Disability Index | 2 weeks (or at day of hospital discharge), 3 months, 12 and 12 months postoperatively
  To observe the change of Oswestry Disability Index as compared to baseline through follow-up terms (min - 0 - the best result, patient is active; max - 50 - the worst result, patient is not physically active)
Change from baseline in The Health Transition Item from SF-36 | 2 weeks (or at day of hospital discharge), 3 months, 12 and 12 months postoperatively
  To observe the The Health Transition Item as compared to baseline through follow-up terms (Patient's answers range from ''Much Better,'' ''Somewhat Better,'' ''About the Same,'' ''Somewhat Worse,'' to ''Much Worse.'')
Change from baseline in lumbar balance parameters | 3 months and 12 months postoperatively
  To observe the change from baseline in segmental lordosis at operated level by full body X-Ray, in degrees
Change from baseline in lumbar balance parameters | 3 months and 12 months postoperatively
  To observe the change from baseline in low lumbar lordosis (L4-S1) by full body X-Ray, in degrees
Change from baseline in lumbar balance parameters | 3 months and 12 months postoperatively
  To observe the change from baseline in sagittal vertical axis by full body X-Ray, in degrees
Change from baseline in lumbar balance parameters | 3 months and 12 months postoperatively
  To observe the change from baseline in full balance integrated index by full body X-Ray, in degrees
Change from baseline in lumbar balance parameters | 12 months postoperatively
  To observe the interbody fusion grade by CT , grades by Tan
Adverse Events | during study, an average of 12 months
  Document Adverse Events (incl. adverse events related to device) occurrence throughout the study

CONTACTS AND LOCATIONS:
Locations (1):
- Priorov National Medical Research Center of Traumatology and Orthopedics, Moscow, Russia